CLINICAL TRIAL: NCT05442268
Title: Duloxetine for Post Operative Analgesia After Modified Radical Mastectomy:A Randomized Controlled Study
Brief Title: Duloxetine for Postoperative Analgesia After Modified Radical Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Abdel monem Elfeky, Principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35146/12/21
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Modified Radical Mastectomy; Postoperative Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen group (Experimental): patients will receive intravenous 500 mg acetaminophen(every 6 hours postoperatively.
  Interventions: Procedure: Acetaminophen group
- Duloxetine group (Experimental): Patients will receive duloxetine 30 mg every 12 hours for 3 days before surgery, 30 mg 2 hours preoperatively and 30 mg 12 hours postoperatively and intravenous 500 mg acetaminophen (every 6 hours postoperatively)
  Interventions: Procedure: Duloxetine group

INTERVENTIONS:
Procedure: Acetaminophen group — patients will receive intravenous 500 mg acetaminophen(every 6 hours postoperatively
  Arms: Acetaminophen group
Procedure: Duloxetine group — Patients will receive duloxetine 30 mg every 12 hours for 3 days before surgery, 30 mg 2 hours preoperatively and 30 mg 12 hours postoperatively and intravenous 500 mg acetaminophen every 6 hours postoperatively
  Arms: Duloxetine group

SUMMARY:
The aim of this study is to evaluate the role of duloxetine in controlling pain after radical mastectomy.

DETAILED DESCRIPTION:
Inadequate control of postoperative pain is associated with increased length of hospital stay, increased hospital cost, sleep disturbance, depression, functional impairment and affects the quality of life.

Modified is one of the commonly performed procedures which is associated with severe postoperative pain.

Preemptive analgesia is the analgesic treatment initiated before the surgical procedure to prevent central sensitization from the noxious stimuli. Drugs such as gabapentin, pregabalin, serotonin-norepinephrine reuptake inhibitors, dexamethasone, and cyclooxygenase-2 inhibitors have been used for preemptive analgesia.

There are contrary results about the role of duloxetine in mangement of acute postoperative pain.

Arecent meta-analysis was done in 2020 that concluded that the currently available evidence does not support the clinical use of duloxetine for the management of acute postoperative pain,so we will discuss that in this study.

There are many studies that have shown that perioperative use of duloxetine for a few days has a significant effect on reducing postoperative pain and analgesic requirements.

Duloxetine is a dual anti-depressant drug that inhibits the neuronal reuptake of serotonin (5-HT) and norepinephrine (NE) modulating the descending inhibitory pain pathways by increasing the availability of serotonin and norepinephrine. Duloxetine is an approved drug for the treatment of post-traumatic depression, major depression, and generalized anxiety disorder. It is also approved for the treatment of various chronic painful syndromes, including neuropathic pain associated with diabetes, chronic musculoskeletal pain, and fibromyalgia.

The mechanisms of action so far described suggest that duloxetine may be useful as an adjunct in the treatment of acute postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients aged (18 - 60) years undergoing modified radical mastectomy. American Society of Anesthesiologists Classification I-II-III

Exclusion Criteria:

Known Allergies to duloxetine.

* Abnormal liver or renal function tests.
* Narrow angle glaucoma.
* Being a chronic opioid abuser (more than 3 months)
* Being on chronic gabapentin or pregabalin (more than 3 months)
* Being on Monoamine oxidase inhibitor, tricyclic antidepressant, or fluvoxamine.
* Pregnant female
* Patients with psychiatric disorders or seizure disorders.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 48 hours postoperatively
  Postoperative Total morphine consumption will be recorded

SECONDARY OUTCOMES:
First analgesic request | 24 hours postoperatively
  First analgesic request will be recorded
Post-operative pain | 48 hours postoperatively.
  Post-operative pain will be assessed by visual analogue score (VAS) from 0-10 scale 0 (no pain) to 10 (the worst imaginable pain) at 2,4,6 h then every 6h
Heart rate | 48 hours postoperatively
  Heart rate will be measured every 30 minutes intraoperative and at 0 hour (direct postoperative) at post anesthesia care unit then at 2,4,6 hours at ward then every 6 hours for 48 hours postoperatively
Mean arterial blood pressure | 48 hours postoperatively
  Mean arterial blood pressure will be measured every 30 minutes intraoperative and at 0 hour (direct postoperative) at post anesthesia care unit then at 2,4,6 hours at ward then every 6 hours for 48 hours postoperatively
Adverse effects | 48 hours postoperatively
  Hypotension, Bradycardia, nausea, dry mouth,diarrhea, constipation,insomnia, somnolence, fatigue, hyperhidrosis and pruritus will be observed and treated accordingly

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University hospitals, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: one year after the end of the study